CLINICAL TRIAL: NCT02470741
Title: Pilot of Letrozole for Uterine Myomas
Acronym: PLUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-15678
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Leiomyoma; Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole (Experimental): Oral letrozole 2.5mg/day
  Interventions: Drug: Letrozole
- Placebo and Letrozole (Placebo Comparator): Intermittent oral letrozole 2.5mg/day for 2 months and an identical placebo capsule for 4 months
  Interventions: Drug: Letrozole; Other: Placebo

INTERVENTIONS:
Drug: Letrozole
  Other Names: Femara
Other: Placebo
  Arms: Placebo and Letrozole

SUMMARY:
PLUM evaluates the drug letrozole as a treatment for uterine fibroids. This study is a randomized, blinded, placebo-controlled trial of oral letrozole among premenopausal women with symptomatic uterine fibroids. Participants will be randomly assigned in a 1:1 ratio to either oral letrozole 2.5mg/day for 6 months (Group A) or intermittent dosing with letrozole 2.5mg/day and an identical placebo capsule (Group B).

ELIGIBILITY:
Inclusion Criteria:

1. ≥21 years old
2. Premenopausal (at least one menses in last 3 months)
3. Symptomatic fibroids (fibroids visualized on ultrasound or MRI and heavy uterine bleeding, pelvic pressure or discomfort, urinary or bowel abnormalities, dyspareunia)
4. Fibroids that are ≤4 in total number or Fibroids that are ≤7 in total number if all fibroids are less than 4cm (40 mm) each
5. Fibroids that are ≤7cm in maximum diameter, on screening imaging, if ≤4 fibroids in total number(fibroid is defined as any mass with radiographic characteristics of fibroid >2cm)
6. Up to date in Pap smear screening and surveillance
7. Endometrial biopsy (required if age>45 years with irregular bleeding) does not indicate premalignant or malignant cells
8. Agree to use non-hormonal barrier method of contraception during study period if at risk for pregnancy
9. Has primary care provider or gynecologist
10. Agrees not to start new medications/treatments for fibroids during the study
11. Able to give informed consent

Exclusion Criteria:

1. Fibroids treated by surgery, radiologic procedure, or GnRH agonist or antagonist in the last 3 months
2. Any submucosal fibroid ≥2cm that is >50% in uterine cavity (FIGO Type 0 or Type 1 fibroids) amenable to hysteroscopic resection
3. Use of exogenous estrogen and/or progestin in the last month. (for 3 month long-acting depoprovera injection, no use in last 3 months)
4. Pregnant, lactating, or planning to become pregnant in the next 6 months
5. Hematocrit <27% or visit to emergency room or hospitalization for fibroid symptoms in the last 3 months (cannot be safely randomized to a placebo)
6. History of osteopenia or osteoporosis
7. History of hyperlipidemia
8. Current liver or kidney disease
9. Unable or unwilling to attend 4 study visits
10. Pelvic imaging concerning for gynecologic cancer or cancer of the genitourinary or gastrointestinal system
11. Does not have primary care provider or gynecologist

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: Fibroid Trials at UCSF — https://clinicaltrials.ucsf.edu/fibroids

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Letrozole | Placebo and Letrozole
Started | 6 | 6
Completed | 3 | 4
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Placebo and Letrozole | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.33 (4.2) | 39.50 (7.4) | 42.92 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 2 | 2 | 4
  Black or African American | 0 | 2 | 2
  Hispanic or Latina | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian/Alaska Native | 0 | 0 | 0
  Other | 1 | 1 | 2
  More than one race reported | 2 | 0 | 2
UFS-QOL Symptom Severity Score [Mean (Standard Deviation); unit: units on a scale] — The Uterine Fibroid Sympton and Quality of Life (UFS-QoL) Symptom Severity score measures self-reported severity of fibroid-related symptoms. Symptoms include: fatigue, sleep, self-image, mood disturbances/psychologic distress, fear of embarrassment, interference with daily activities, relationships with family and friends, and sexual functioning.
  Scores range from 0 to 100; higher scores indicate greater symptom severity.
  units on a scale | 53.65 (25.00) | 42.71 (9.0) | 48.18 (18.8)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Fibroid-related Symptoms After Treatment With Letrozole
Description: The Uterine Fibroid Sympton and Quality of Life (UFS-QoL) Symptom Severity score measures self-reported severity of fibroid-related symptoms. Symptoms include: fatigue, sleep, self-image, mood disturbances/psychologic distress, fear of embarrassment, interference with daily activities, relationships with family and friends, and sexual functioning.
  Scores range from 0 to 100; higher scores indicate greater symptom severity.
Time Frame: Baseline to 2 Months
Population: The final analysis excludes one participant in the placebo/letrozole group who dropped out of the study after baseline but prior to starting study medication and the Month 2 visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Letrozole | Placebo and Letrozole
Number analyzed (Participants) | 6 | 5
units on a scale | -10.42 [-24.63 to 3.97] | 1.43 [-14.14 to 16.99]
Statistical Analysis 1: Comparison: Letrozole vs Placebo and Letrozole; Null hypotheses: Letrozole is not associated with an improvement in the UFSQOL Overall Score; Test type: Superiority; p = 0.24, Mixed Models Analysis; Repeated measures mixed models, with unstructured co-variance matrix; Mean Difference (Net) = -11.85, 95% CI 2-sided [-32.92 to 9.23] — Model generated LS Mean Differences

ADVERSE EVENTS:
Time Frame: 7 months. Adverse Events were collected beginning at Baseline until 1 month after study completion.
Arm/Group | Letrozole | Placebo and Letrozole
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=6) | Placebo and Letrozole (N=6)
Dizziness/Light-headedness (General disorders) | 1 (1) | 0 (0)
Pelvic pressure increasing urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Bleeding between periods (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Irritable (Psychiatric disorders) | 0 (0) | 1 (1)
Pain in uterus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oily skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flashes/night sweats (Vascular disorders) | 0 (0) | 1 (1)
Stomach aches (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle or joint pain/strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT02470741/Prot_SAP_000.pdf